CLINICAL TRIAL: NCT06719466
Title: the Effect of Diet Intervention on Obesity
Brief Title: Diet Intervention on Obesity Related Complication
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Manna (Other)
Responsible Party: Sponsor-Investigator, Zhang Manna, professor, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20240624
Record Dates: First submitted 2024-06-23; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Obese; Stomach Diseases
MeSH Terms: conditions — Obesity; Stomach Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- linoleic acid (LA) (Experimental): diet intervention（diet guidance with low linoleic acid (LA) ）
  Interventions: Other: low linoleic acid (LA)

INTERVENTIONS:
Other: low linoleic acid (LA) — diet guidance with low linoleic acid (LA) diet

SUMMARY:
Obesity has become a global epidemic, with more than 4 billion people expected to be overweight/obese by 2035, accounting for more than half of the world's population. Currently, there are sixteen recognized complications directly related to obesity, including gastroesophageal reflux disease. In recent years, people have increasingly paid attention to the damage caused by obesity to the stomach. In addition to gastroesophageal reflux disease, obesity also leads to various forms of gastric mucosal damage related diseases, such as gastric ulcers, chronic gastritis, intestinal metaplasia, and so on. This stuty aimed to observe the diet intervention on obesity related stomach.

DETAILED DESCRIPTION:
Western foods high in fat, sugar, fiber and additives can lead to a series of health problems, ultimately leading to obesity and obesity-related complications. The gastrointestinal tract is directly connected to the outside world, so its influence on dietary factors cannot be underestimated. In recent years, the intake of ω-6 polyunsaturated fatty acids (ω-6 PUFAs) in the Western diet is 10-20 times higher than the normal range, of which the seriously excessive linoleic acid (LA) is also getting more and more attention

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent before carrying out any trial-related activity, which is any procedure carried out as part of a trial, including the identification of activities suitable for the trial
2. Men and premenopausal women, ages 18-65 at the time of signing the informed consent form
3. Obese patients are diagnosed based on a body mass index (BMI) of 28-40kg/m2

Exclusion Criteria:

1）Patients who do not possess or lose the ability to make their judgment, are unable to understand the purpose of the study, or are unwilling to cooperate with it; 2) Heart, liver, kidney dysfunction，and systemic diseases, such as various malignant tumors, systemic allergic diseases, and autoimmune diseases; 3）Drug or alcohol dependence, intellectual disability, mental disorders; 4）Pregnant and lactating women; 5) Confirmed Helicobacter pylori infection (PPI, bismuth, and antibiotics were stopped for at least 4 weeks, and any of the following tests were positive: non-invasive HP test such as urea breath test, monoclonal stool Helicobacter pylori antigen test, serum soluble Helicobacter pylori antigen test; Invasive Hp test included rapid urease test and tissue section staining); 6）diagnosis of acute gastric mucosal lesions; 7）the patient was diagnosed with chronic gastritis according to the new Sydney system visual simulation scoring method and the pathological diagnostic criteria of chronic gastritis in China; 8） histological and imaging examinations, adenocarcinoma was diagnosed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
body weight | 12 weeks
  stomach injury scale

SECONDARY OUTCOMES:
metabolic markers | 12 weeks
  change in body weight and metabolic markers

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, China

DOCUMENTS (2):
  • Study Protocol (2024-06-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT06719466/Prot_000.pdf
  • Informed Consent Form (2024-06-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT06719466/ICF_001.pdf